CLINICAL TRIAL: NCT02760693
Title: SPICS (Secure Platform for Integrating Clinical Studies) for Recurrent (Bipolar) Affective Disorders for Long Term Follow up Treatment Regiments and Outcome in a Natural Setting
Brief Title: Bipolar Cohort Neunkirchen, Final Statement
Status: Completed | Type: Observational
Sponsor: Österreichische Gesellschaft für Bipolare Erkrankungen (Other)
Responsible Party: Sponsor
Other Study IDs: Protocoll2; SPICS2010-2 (Other: Österreichische Gesellschaft für Bipolare Erkrankungen); NCT01792128 (obsolete NCT alias)
Record Dates: First submitted 2016-04-27; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-04

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder, naturalistic cohort study,; defined catchment area,long term treatment
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- bipolar patients: unselected admissions of bipolar patients

SUMMARY:
monitoring system and data base for long term follow up of various treatment strategies in a naturalistic setting of recurrent affective disorders (unipolar, bipolar) open study design, prospective & retrospective

DETAILED DESCRIPTION:
all hospitalized patients of a defined mixed urban and more rural area were consecutively interviewed at admission and entered into the data base. at discharge they gave written informed consent for further tracking and interviews.

ELIGIBILITY:
Inclusion Criteria:

* bipolar

Exclusion Criteria:

* all other diagnoses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community of wiener neustadt and neunkirchen
Sampling Method: Non-Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2000-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
relapses, hospital admissions, number of participants with adverse events as a measure of safety and tolerability | patients from the cohort are contacted once a year (1 to 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Christian A. Simhandl, Principal Investigator — Bipolar Zentrum WN
Locations (1):
- BIPOLAR Zentrum Wiener Neustadt, Wiener Neustadt, Lower Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simhandl C, Radua J, Konig B, Amann BL. The prevalence and effect of life events in 222 bipolar I and II patients: a prospective, naturalistic 4 year follow-up study. J Affect Disord. 2015 Jan 1;170:166-71. doi: 10.1016/j.jad.2014.08.043. Epub 2014 Sep 6. PMID 25240845
- [Background] Simhandl C, Radua J, Konig B, Amann BL. Prevalence and impact of comorbid alcohol use disorder in bipolar disorder: A prospective follow-up study. Aust N Z J Psychiatry. 2016 Apr;50(4):345-51. doi: 10.1177/0004867415585855. Epub 2015 May 13. PMID 25972409
- [Result] Simhandl C, Konig B, Amann BL. A prospective 4-year naturalistic follow-up of treatment and outcome of 300 bipolar I and II patients. J Clin Psychiatry. 2014 Mar;75(3):254-62; quiz 263. doi: 10.4088/JCP.13m08601. PMID 24717379